CLINICAL TRIAL: NCT06097338
Title: Quantitative US for Evaluation of Hepatic Steatosis in MAFLD With UDFF
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QFS-UDFF2023
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Fatty Liver Disease, Nonalcoholic
Keywords: metabolism related fatty liver disease (MAFLD); Ultrasound Derived Fat Fraction (UDFF); bariatric surgery; Shear wave elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MAFLD patients: MAFLD patients undergoing weight loss surgery
  Interventions: Procedure: bariatric surgery (BS)
- healthy volunteers: healthy volunteers

INTERVENTIONS:
Procedure: bariatric surgery (BS) — bariatric surgery (BS) is a very attractive choice for severely obese patients. After bariatric surgery, long-term weight loss (15%-25%) and diabetes remission can occur [16], as well as long-term mortality, cardiovascular events and tumor occurrence [17]. Regardless of the surgical procedure used for weight loss surgery, studies have shown that weight loss surgery can significantly reduce the liver NAFLD activity score (from 5 to 1), and 33.8% of patients have reduced liver fibrosis [18]. The follow-up results for a longer period of time (10 years) also indicate that weight loss surgery significantly reduces the occurrence of major adverse outcomes related to liver cirrhosis, liver cancer, liver transplantation, and liver related deaths
  Groups: MAFLD patients

SUMMARY:
Ultrasound Derived Fat Fraction (UDFF) Evaluation of Metabolic Related Fatty Liver Disease (MAFLD) in obesity Patients Metabolic fatty liver disease (MAFLD), formerly known as Nonalcoholic Fatty Liver Disease (NAFLD), is the most common chronic liver disease in the world at present, with a incidence rate of about 30%. In the United States, NAFLD is the third leading cause of hepatocellular carcinoma, and early assessment and diagnosis of liver steatosis characteristics are crucial for timely treatment or intervention to reduce the risk of liver fibrosis and inhibit disease progression. Liver biopsy is considered as the "gold standard" for evaluating, grading, and determining inflammatory activity of liver steatosis and fibrosis. However, liver biopsy are invasive and pathological evaluation differences among observers, which makes it difficult to widely use and repeat, especially for dynamic evaluation of patients during the treatment process.

Ultrasound Derviced Fat Fraction (UDFF) is a unique technology for non-invasive quantification of liver fat content, which is equipped on the Siemens ACUSON Sequoia ultrasound system. UDFF is calculated from two parameter values: attenuation coefficient (AC) and backscatter coefficient (BSC). SWE (shear wave elastography) is becoming widely used, and is recommended for the evaluation of liver fibrosis by some guidelines in patients with chronic liver diseases, such as viral hepatitis. These two technologies (UDFF+SWE) can be achieved on the same probe, and this detection technology is non-invasive, painless, simple, and reliable.

Bariatric surgery (BS), also known as metabolic weight loss surgery, is currently recognized as the most significant and long-lasting method for treating obesity. It can significantly improve obesity related comorbidities, as well as long-term improvement in postoperative quality of life and mental state.

This study will aim on analysis of the liver ultrasound characteristics of patients who plan to undergo bariatric surgery. By using UDFF and elastic shear wave technology (UDFF+SWE), a new non-invasive ultrasound evaluation method for MAFLD grading diagnosis of simple fatty liver, fatty hepatitis, liver fibrosis, and related cirrhosis will be proposed, and the incidence and risk factors of MAFLD in overweight and obese patients will be explored, The reversal effect of weight loss therapy on MAFLD in obese patients.

DETAILED DESCRIPTION:
1. Research background

MAFLD (NAFLD) is considered to be the most common adult chronic liver disease in the world, affecting more than 30% of the world's population. Previous studies have shown that 55%-80% of NAFLD patients have type 2 diabetes. Early assessment and diagnosis of liver steatosis characteristics is crucial for timely treatment or intervention to reduce the risk of liver fibrosis and inhibit disease progression in MAFLD/NAFLD.

At present, liver biopsy is considered as the "gold standard" for evaluating, grading, and determining inflammatory activity of liver steatosis and fibrosis. However, liver biopsy has certain limitations, such as pain, bleeding, infection, bile leakage, leading to the inability to widely use and repeat detection of liver biopsy, especially for dynamic evaluation of patients during treatment .

Therefore, in recent years, non-invasive diagnosis of liver fat content has attracted much attention. Conventional ultrasound is the most commonly used imaging method for evaluating liver steatosis. Conventional abdominal CT can also be used to diagnose fatty liver, but its sensitivity is similar to or even lower than ultrasound, accompanied by radiation, which limits its application in screening and evaluation of fatty liver. Other imaging methods include magnetic resonance spectroscopy (MRS) and magnetic resonance chemical shift coding (MRI) . Magnetic resonance spectroscopy (MRS) uses the difference in resonance frequency between water and fat proton signals to measure proton density fat fraction (PDFF). MRI-PDFF is closely related to histological evaluation of liver fat content and is currently the most sensitive non-invasive method for detecting and quantifying liver steatosis.

UDFF is a novel and unique technology for non-invasive quantification of liver fat content, equipped on the Siemens ACUSON Sequoia ultrasound system. UDFF is calculated from two parameter values: Attenuation Coefficients (AC) and Backscatter Coefficients (BSC). These two parameters are determined by comparing the frequency content of backscattered echo signals at different depths within the tissue and the reference module of the simulated tissue. The AC and BSC values of the reference module are known to be fixed. By comparing, the attenuation of tissues can be separated and their AC can be estimated. The ratio of two spectra and the AC of the module can also be used to estimate the backscatter coefficient of tissue samples. After calculating and estimating the BSC, a unique proprietary mathematical algorithm was used to estimate the UDFF value of the tissue sample at 3MHz. Convert BSC to UDFF in percentage using a special algorithm (P) (linearize the 3MHz BSC to obtain UDFF). Unlike AC and BSC values, the UDFF obtained through special algorithms has a linear relationship with liver fat content. As the fat content level increases, the UDFF index value also increases.

UDFF can quickly and non-invasive quantify liver fat content within seconds during routine abdominal ultrasound examination. This technology is non-invasive, painless, simple, and reliable, and will contribute to the diagnosis and dynamic evaluation of MAFLD during the treatment process, playing an important role in the patient's prognosis.

In addition to fat deposition in the liver (balloon like transformation of liver cells), liver fibrosis is an important monitoring indicator for the progression of MAFLD. On the Siemens Sequoia ultrasound system, the measurement of shear wave elastography (SWE) can be achieved on the same probe as UDFF technology, simultaneously.

As MAFLD is a series of diseases, and may be combined with a variety of metabolic related complications, such as cardiovascular disease, type 2 diabetes, leading to the complexity of MAFLD treatment. The initial treatment plan for MAFLD currently involves lifestyle changes, including controlling diet and exercise, ultimately achieving weight loss. Weight loss, regardless of the method used, is strongly correlated with histological improvement in MAFLD, with even a 5% weight loss indicating a reduction in patients' fatty liver.

Bariatric surgery (BS) is a very attractive choice for severely obese patients. After bariatric surgery, long-term weight loss (15%-25%) and diabetes remission can occur, as well as mortality, cardiovascular events and tumor occurrence. Studies have shown that bariatric surgery can significantly reduce the liver NAFLD activity score (from 5 to 1), and 33.8% of patients have reduced liver fibrosis. Due to the use of liver biopsy to evaluate liver histological changes in NAFLD/MAFLD observation during bariatric surgery, liver biopsy cannot be widely used and repeatedly detected due to its invasive nature and differences in pathological evaluation among observers. Especially for patients during treatment and follow-up, flexible dynamic evaluation is difficult to achieve.

This study will conduct a detailed analysis of the liver ultrasound characteristics of patients who plan to undergo bariatric surgery. By using UDFF+SWE technology, a new method for non-invasive evaluation of MAFLD grading diagnosis of simple fatty liver, fatty hepatitis, fatty liver fibrosis, and related cirrhosis will be proposed. The incidence and risk factors of overweight and obese patients with MAFLD will be explored, and the reversal effect of weight loss treatment on MAFLD in obese patients will be explored.

2 Research aims

The aim of this study is to prospectively evaluate UDFF for detection of hepatic steatosis and quantification of liver fat content, meanwhile to assess SWE for detection of liver fibrosis using a DAX probe in patients who plan to undergo bariatric surgery. Through UDFF technology and elastic shear wave technology, a new non-invasive ultrasound evaluation method for MAFLD grading diagnosis of simple fatty liver, fatty hepatitis, fatty liver fibrosis, and related cirrhosis will be proposed.

3 Research protocol

UDFF technology was used to detect liver fat fraction in patients who plan to undergo bariatric surgery, while SWE was used to monitor liver stiffness. Pathological diagnosis was used as the gold standard to determine the correlation between relevant feature quantities and fibrosis, inflammation grading, and steatosis grading. Multiple regression equations were established to form UDFF scores for different degrees of MAFLD and different grading diagnostic thresholds. Analyze its diagnostic effectiveness through internal and external verification methods.

Each participant will undergo ultrasound examination (UDFF+ SWE) before bariatric surgery and 1 month, 3 months, 6 months and 12months after surgery.

3.1 Observe items

3.1.1 General clinical information collection

Gender, age, height, weight, waist, BMI, blood pressure, history of hepatitis, history of diabetes, antiviral treatment.

Alcohol drinking history (calculation formula: daily alcohol intake (grams)=alcohol consumption (milliliters) × Alcohol content (%) × Specific gravity of alcohol (0.8)

3.1.2 Serum biochemical parameters 3.1.2.1 Blood testing: RBC (red blood cells), HGB (hemoglobin), WBC (white blood cells) NEUT% (neutrophil percentage), PLT (platelet count); 3.1.2.2 Serum TB (total bilirubin), DB (direct bilirubin), IB (indirect bilirubin), ALB (albumin), AST (aspartate aminotransferase), ALT (alanine aminotransferase), GGT（ γ- Glutamyl transpeptidase, ALP (alkaline phosphatase); SCr (blood creatinine), UA (blood uric acid); TG (triglycerides), CHOL (total cholesterol), HDL-C (high-density lipoprotein cholesterol), LDL-C (low-density lipoprotein cholesterol); glucose,insulin, GHb (glycated hemoglobin); 3.1.2.3 Blood coagulation test : PT (prothrombin time), INR (international standardized ratio); Interleukin 6/8, CRP (C-reactive protein); 3.1.2.4 Serum HBsAg、HBsAb、HBeAg、HBeAb、HBcAb、HBV DNA 3.1.3 Conventional ultrasound and UDFF+SWE examination: 3.1.3.1 Equipment: Siemens ACUSON Sequoia ultrasound system with C5-1 probe and DAX probe.

3.1.3.2 Preparation before examination: patients fast for at least 4 hours and after resting for at least 20 minutes. Avoid testing after diet (especially caffeine) and smoking.

3.1.3.3 UDFF observer training: It should be performed by an experienced sonographer. Provide more than 50 training sessions for beginners.

3.1.3.4 Instrument settings: Unified settings for frequency, gain, etc. The total depth of the image during UDFF measurement is within 15cm.

3.1.3.5 Conventional ultrasound examination (C5-1 probe): abdominal wall thickness; parenchymal echo of the liver and spleen; size of spleen; size of liver lobes: Smooth degree of liver capsule; Portal vein diameter and blood flow velocity.

3.1.3.6 UDFF+SWE examination (DAX probe): The participant lay in a supine position, with the probe placed between the right ribs or under the xiphoid process, avoiding the intrahepatic duct structure. The sampling boxes are placed in the right lobe of the liver (S5 best, followed by S8) and the left lobe of the liver (S2 or S3 segment), respectively. Instruct the participant to calm down and hold their breath before measuring to avoid Valsalva movements. Measure the left and right lobes of the liver 5 times, store the map and record the measured values.

3.1.3.7 Images Storages: 3.1.3.7.1 Liver grayscale images left lobes: longitudinal and transverse sections under the xiphoid process (including the smoothness of the liver capsule); right lobe: oblique diameter under the right rib (showing the second hepatic hilum), right intercostal section, and liver kidney contrast section; 3.1.3.7.2 Portal vein diameter, color Doppler ultrasound, and flow velocity measurement maps.

3.1.3.7.3 Measurement and storage of abdominal wall thickness; 3.1.3.7.4 Measurement of spleen length and thickness. 3.1.3.7.5 UDFF+SWE: 5 measurement pictures for each left and right lobes

3.1.4 Pathological examination (before surgery): Using 18g or 20g puncture needles for ultrasound-guided percutaneous liver biopsy, the length of the tissue specimen should be≥ 15mm and include at least 6 complete portal areas. All liver biopsy specimens were independently evaluated by senior pathologists who were unaware of clinical data. The liver Steatosis, Activity, and Fibrosis (SAF) scoring system will be used as pathological diagnosis standard for MAFLD diagnosis.

3.2 Statistical Analysis Plan

3.2.1 Descriptive statistics on demographic data will be presented as total number and percentage. Continuous and normally distributed data will be analyzed with ANOVA and reported as mean and SD. Continuous and not normally distributed data will be analyzed using the Kruskal-Wallis test and reported as median and interquartile ranges (IQR). For categoric data, variables will be described as number and percentage, and the Fisher exact test is used for analysis.

3.2.2 The cut-off value for the diagnosis of hepatic steatosis was 5% both for UDFF, as determined by previous studies. Agreement and correlation between UDFF and pathological liver steatosis will be evaluated by the Bland-Altman dierence plot, one-sample T test, and Pearson's correlation test. The diagnostic value of B-mode US and UDFF measurements for the detection of steatosis will be assessed by the calculation of sensitivity, specificity, positive and negative predictive values (PPV and NPV), and accuracy. Receiver operating characteristic curves (ROCs) will be constructed for B-mode US and UDFF by taking pathological liver steatosis the standard of reference, and area under the curves (AUC-ROC) will be calculated; comparison of ROC curves will be performed with the method described by Delong et al. p values ≤ 0.05 will be considered statistically significant. Statistical analysis will be performed using commercially available software (SPSS 23, IBM; and MedCalc 17.9, MedCalc Software).

ELIGIBILITY:
Inclusion Criteria:

1. Chinese citizens aged 18 ≤ 85;
2. Routine ultrasound reveals diffuse or non-uniform fatty liver disease in the liver;
3. Conform to the MAFLD diagnostic criteria issued by the international guidelines: histological (liver biopsy), imaging or blood biomarker evidence based on liver fat accumulation (hepatocyte steatosis), and combine one of the following three conditions: overweight/obesity (BMI ≥ 23 kg/m2), type 2 diabetes, and metabolic dysfunction. The definition of metabolic dysfunction is the presence of at least two of the following metabolic risk factors: 1. waist circumference (for Asians) ≥ 90/80 cm (male/female);2. Arterial blood pressure ≥ 130/85 mmHg is being treated with antihypertensive drugs; 3. Hypertriglyceridemia (TG): fasting serum TG ≥ 150 mg/dl (≥ 1.70 mmol/L) or being treated with lipid-lowering drugs; 4. High density lipoprotein cholesterol (HDL-c) emia: fasting serum HDL-c<40 mg/dl (<1.0 mmol/L) for males,<50 mg/dl (<1.3 mmol/L) for females, or specific medication treatment;5. Pre diabetes (i.e. fasting blood glucose level 100-125 mg/dl [5.6-6.9 mmol/L], or blood glucose level 140-199 mg/dl [7.8-11.0 mmol] 2 hours after meal or HbA1c 5.7% -6.4% [39-47 mmol/mol]);6. Steady state model evaluation of insulin resistance score ≥ 2.5;7. Plasma C-reactive protein levels>2 mg/L.
4. Those who plan to undergo liver histopathological diagnosis or MRI-PDFF assessment of the degree of fatty liver within one week;
5. No significant risk of bleeding (platelet ≥ 50x109/L, international standardized ratio of prothrombin time INR ≤ 1.5);
6. The patient agrees to join this study and signs an informed consent form.

Exclusion Criteria:

* 1. No histopathological diagnosis or MRI-PDFF was found;
* 2. The interval between the ultrasound UDFF examination and the histopathological examination or MRI-PDFF examination is more than one week;
* 3. Pregnancy;
* 4. Incomplete medical history information.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the hospitalized patients plan to undergo bariatric surgery in the First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The combined detection of UDFF and SWE based on ultrasound images | 12 months
  UDFF technology will be used to detect liver fat content in patients who plan to undergo weight loss surgery, while SWE will be used to monitor liver hardness. Pathological diagnosis will be used as the gold standard to determine the correlation between relevant feature quantities and fibrosis grade, inflammation grade grade, and lipid degeneration grade. Multiple regression equations will be established to form UDFF scores for different degrees of MAFLD and different grading diagnostic thresholds. Analyze its diagnostic effectiveness through internal and external verification methods.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Ma, MD，PHD, Study Director — Department of Ultrasound, Shandong Provincial Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aminian A, Al-Kurd A, Wilson R, Bena J, Fayazzadeh H, Singh T, Albaugh VL, Shariff FU, Rodriguez NA, Jin J, Brethauer SA, Dasarathy S, Alkhouri N, Schauer PR, McCullough AJ, Nissen SE. Association of Bariatric Surgery With Major Adverse Liver and Cardiovascular Outcomes in Patients With Biopsy-Proven Nonalcoholic Steatohepatitis. JAMA. 2021 Nov 23;326(20):2031-2042. doi: 10.1001/jama.2021.19569. PMID 34762106
- [Background] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783
- [Background] Bouchard P, Al-Masrouri S, Demyttenaere S, Court O, Andalib A. Long-term Impact of Bariatric Surgery on Major Adverse Cardiovascular Events in Patients with Obesity, Diabetes and Hypertension: a Population-level Study. Obes Surg. 2022 Mar;32(3):771-778. doi: 10.1007/s11695-021-05849-1. Epub 2022 Jan 21. PMID 35060016
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Aminian A, Brethauer SA, Navaneethan SD, Singh RP, Pothier CE, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric Surgery versus Intensive Medical Therapy for Diabetes - 5-Year Outcomes. N Engl J Med. 2017 Feb 16;376(7):641-651. doi: 10.1056/NEJMoa1600869. PMID 28199805
- [Background] Ferraioli G, Filice C, Castera L, Choi BI, Sporea I, Wilson SR, Cosgrove D, Dietrich CF, Amy D, Bamber JC, Barr R, Chou YH, Ding H, Farrokh A, Friedrich-Rust M, Hall TJ, Nakashima K, Nightingale KR, Palmeri ML, Schafer F, Shiina T, Suzuki S, Kudo M. WFUMB guidelines and recommendations for clinical use of ultrasound elastography: Part 3: liver. Ultrasound Med Biol. 2015 May;41(5):1161-79. doi: 10.1016/j.ultrasmedbio.2015.03.007. Epub 2015 Mar 20. PMID 25800942
- [Background] Ferraioli G, Wong VW, Castera L, Berzigotti A, Sporea I, Dietrich CF, Choi BI, Wilson SR, Kudo M, Barr RG. Liver Ultrasound Elastography: An Update to the World Federation for Ultrasound in Medicine and Biology Guidelines and Recommendations. Ultrasound Med Biol. 2018 Dec;44(12):2419-2440. doi: 10.1016/j.ultrasmedbio.2018.07.008. Epub 2018 Sep 9. PMID 30209008
- [Background] Labyed Y, Milkowski A. Novel Method for Ultrasound-Derived Fat Fraction Using an Integrated Phantom. J Ultrasound Med. 2020 Dec;39(12):2427-2438. doi: 10.1002/jum.15364. Epub 2020 Jun 11. PMID 32525261
- [Background] Ferraioli G, Kumar V, Ozturk A, Nam K, de Korte CL, Barr RG. US Attenuation for Liver Fat Quantification: An AIUM-RSNA QIBA Pulse-Echo Quantitative Ultrasound Initiative. Radiology. 2022 Mar;302(3):495-506. doi: 10.1148/radiol.210736. Epub 2022 Jan 25. PMID 35076304
- [Background] Kim M, Kang BK, Jun DW. Comparison of conventional sonographic signs and magnetic resonance imaging proton density fat fraction for assessment of hepatic steatosis. Sci Rep. 2018 May 17;8(1):7759. doi: 10.1038/s41598-018-26019-x. PMID 29773823
- [Background] Palmeri ML, Milkowski A, Barr R, Carson P, Couade M, Chen J, Chen S, Dhyani M, Ehman R, Garra B, Gee A, Guenette G, Hah Z, Lynch T, Macdonald M, Managuli R, Miette V, Nightingale KR, Obuchowski N, Rouze NC, Morris DC, Fielding S, Deng Y, Chan D, Choudhury K, Yang S, Samir AE, Shamdasani V, Urban M, Wear K, Xie H, Ozturk A, Qiang B, Song P, McAleavey S, Rosenzweig S, Wang M, Okamura Y, McLaughlin G, Chen Y, Napolitano D, Carlson L, Erpelding T, Hall TJ. Radiological Society of North America/Quantitative Imaging Biomarker Alliance Shear Wave Speed Bias Quantification in Elastic and Viscoelastic Phantoms. J Ultrasound Med. 2021 Mar;40(3):569-581. doi: 10.1002/jum.15609. Epub 2021 Jan 7. PMID 33410183
- [Background] Osawa H, Mori Y. Sonographic diagnosis of fatty liver using a histogram technique that compares liver and renal cortical echo amplitudes. J Clin Ultrasound. 1996 Jan;24(1):25-9. doi: 10.1002/(SICI)1097-0096(199601)24:13.0.CO;2-N. PMID 8655663
- [Background] Pai RK, Kleiner DE, Hart J, Adeyi OA, Clouston AD, Behling CA, Jain D, Kakar S, Brahmania M, Burgart L, Batts KP, Valasek MA, Torbenson MS, Guindi M, Wang HL, Ajmera V, Adams LA, Parker CE, Feagan BG, Loomba R, Jairath V. Standardising the interpretation of liver biopsies in non-alcoholic fatty liver disease clinical trials. Aliment Pharmacol Ther. 2019 Nov;50(10):1100-1111. doi: 10.1111/apt.15503. Epub 2019 Oct 3. PMID 31583739
- [Background] Matteoni CA, Younossi ZM, Gramlich T, Boparai N, Liu YC, McCullough AJ. Nonalcoholic fatty liver disease: a spectrum of clinical and pathological severity. Gastroenterology. 1999 Jun;116(6):1413-9. doi: 10.1016/s0016-5085(99)70506-8. PMID 10348825
- [Background] Sheka AC, Adeyi O, Thompson J, Hameed B, Crawford PA, Ikramuddin S. Nonalcoholic Steatohepatitis: A Review. JAMA. 2020 Mar 24;323(12):1175-1183. doi: 10.1001/jama.2020.2298. PMID 32207804
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Younossi ZM. Non-alcoholic fatty liver disease - A global public health perspective. J Hepatol. 2019 Mar;70(3):531-544. doi: 10.1016/j.jhep.2018.10.033. Epub 2018 Nov 9. PMID 30414863
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630